CLINICAL TRIAL: NCT03647683
Title: Self-Compassion and Acute Pain - an Experimental Investigation
Brief Title: Self-Compassion and Acute Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philipps University Marburg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-60v
Record Dates: First submitted 2018-08-01; First posted 2018-08-27 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Acute Pain
MeSH Terms: conditions — Acute Pain | interventions — Osteogenesis, Distraction

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of three experimental groups in parallel for the duration of the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Self-Compassion (Experimental): After pretreatment heat pain assessment, participants are introduced to the concept of self-compassion. Participants practice the new strategy with heat pain stimuli three times. Next, the posttreatment pain assessment is conducted. For a one week period, participants receive daily self-compassion audio-interventions. Afterwards, the follow-up pain assessment is conducted.
  Interventions: Other: Self-Compassion; Other: Heat pain
- Acceptance (Experimental): After pretreatment heat pain assessment, participants are introduced to the concept of acceptance. Participants practice the new strategy with heat pain stimuli three times. Next, the posttreatment pain assessment is conducted. For a one week period, participants receive daily acceptance audio-interventions. Afterwards, the follow-up pain assessment is conducted.
  Interventions: Other: Acceptance; Other: Heat pain
- Distraction (Experimental): After pretreatment heat pain assessment, participants are introduced to the concept of distraction. Participants practice the new strategy with heat pain stimuli three times. Next, the posttreatment pain assessment is conducted. For a one week period, participants receive daily distraction audio-interventions. Afterwards, the follow-up pain assessment is conducted.
  Interventions: Other: Distraction; Other: Heat pain

INTERVENTIONS:
Other: Self-Compassion — Participants are introduced to the concept of self-compassion. Treating oneself with kindness, while being mindfully aware of the present moment as well as the fact that suffering is part of human life - a shared human experience.
  Participants are instructed to use this strategy to cope with the following heat stimulus.
  Arms: Self-Compassion
Other: Acceptance — Participants are introduced to the concept of acceptance. Thoughts, Emotions and Reactions do not need to be related. Being aware of the present moment helps with accepting the present state and reacting contradictory to the thoughts and feelings.
  Participants are instructed to use this strategy to cope with the following heat stimulus.
  Arms: Acceptance
Other: Distraction — Participants are introduced to the concept of distraction. Distracting oneself from the present situation helps with not perceiving pain, painful thoughts or feelings.
  Participants are instructed to use this strategy to cope with the following heat stimulus.
  Arms: Distraction
Other: Heat pain — Participants receive heat pain stimuli using the Thermo Sensory Analyser (TSA-II), a commonly used device to study pain sensation and analgesic effects.

SUMMARY:
Research on self-compassion suggests its impact in the context of pain. In the current study, the investigators evaluate a short self-compassion intervention for coping with acute pain.

DETAILED DESCRIPTION:
Self-compassion comprises three components: self-kindness, common humanity and mindfulness. Empirical evidence shows the relevance of self-compassion in the context of negative emotions such as depression, anxiety and anger. Research on chronic pain is promising yet limited. Self-compassion is associated with better pain-coping, pain-acceptance and quality of life, as well as reduced pain-related disability and burdening emotions. Experimental investigations on induced pain are missing. The aim of the current study is to evaluate a short self-compassion intervention for pain.

First, a heat stimulus is induced to all participants which is to be tolerated as long as possible and evaluated in intensity and unpleasantness. Next, participants receive a coping-strategy which they are randomly assigned to. Three different strategies are evaluated: (1) self-compassion, treating oneself with kindness while being mindfully aware of the painful stimulus, (2) acceptance, accepting the painful stimulus as well as pain-related thoughts, not trying to change, (3) distraction, distracting oneself from the painful stimulus and trying not to perceive the pain or painful thoughts. Participants practice the strategy with the painful heat stimulus three times. Then, they receive another heat stimulus which is to be tolerated as long as possible and evaluated. During the next week, participants obtain daily practices via e-mail for further fostering of the learned strategy. Finally, participants receive, tolerate and evaluate pain again in the laboratory.

ELIGIBILITY:
Inclusion Criteria:

* sufficient german language knowledge
* at least 18 years old

Exclusion Criteria:

* acute or chronic pain conditions
* drug or pain-medication (last 24 hours)
* Raynaud's disease
* high blood pressure
* neuropathy, coronary diseases
* diabetes, current alcohol
* studying psychology longer than two years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2018-04-15 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Individual heat pain tolerance | Baseline, 45 min, 1 week
  Change in the individual heat pain tolerance (the point when participants cannot stand the heat pain stimulus any longer)

SECONDARY OUTCOMES:
Pain intensity | Baseline, 45 min, 1 week
  Change in subjective pain intensity assessed using a numeric rating scale (ranging from 0 to 10, with higher values reflecting more pain intensity)
Change in pain unpleasantness scale | Baseline, 45 min, 1 week
  Change in subjective pain unpleasentness assessed using a numeric rating scale (ranging from 0 to 10, with higher values reflecting more pain unpleasentness)
Change in self-compassion | Baseline, 45 min, 1 week
  Change in overall self-compassion assessed using the self-compassion scale (Neff, 2003) (higher values indicating higher self-compassion

CONTACTS AND LOCATIONS:
Overall Officials: Anja C Schmitt, Principal Investigator — Philipps University Marburg
Locations (1):
- Philipps-University of Marburg, Marburg, Hesse, Germany

IPD SHARING:
Plan to Share IPD: No